CLINICAL TRIAL: NCT01206283
Title: Modified Lund Concept Versus Cerebral Perfusion Pressure-targeted Therapy: A Randomized Controlled Study in Patients With Secondary Brain Ischaemia.
Brief Title: A Study Comparing Modified Lund Concept and Cerebral Perfusion Pressure-targeted Therapy in Secondary Brain Ischaemia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sarajevo (Other)
Responsible Party: Kemal Dizdarevic, Clinical Center University of Sarajevo, Bosnia and Herzegovina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 030531674
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Brain Injuries; Subarachnoid Hemorrhage
Keywords: traumatic brain injury; subarachnoid hemorrhage; secondary brain ischemia; microdialysis; modified Lund concept; cerebral perfusion pressure; intracranial pressure
MeSH Terms: conditions — Brain Injuries; Subarachnoid Hemorrhage; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cerebral perfusion pressure-targeted (Active Comparator): 15 comatose operated patients after aneurysmal subarachnoid haemorrhage and severe traumatic brain injury respectively were managed postoperatively using cerebral perfusion pressure-targeted therapy according to the American Associations of Neurological Surgeons. Results were categorised into different Glasgow Outcome Scores.
  Interventions: Procedure: Cerebral perfusion pressure-targeted therapy
- Intracranial pressure-targeted therapy (Active Comparator)
  Interventions: Procedure: Modified Lund concept

INTERVENTIONS:
Procedure: Modified Lund concept — After surgical evacuation of intracranial mass lesion and clipping of aneurysm the objectives were achieved:
  * Reduction of cerebral energy metabolism with fentanyl (2-5 µg/kg/h) and thiopenthal (0.5-3 mg/kg/h);
  * Maintenance of colloid osmotic pressure with administration of red cell and albumin/plasma transfusions to maintain Hb/s 125-140 g/L and Alb/s ≈40 g/L;
  * Reduction of capillary hydrostatic pressure with α2-agonist clonidine (0.4-0.8 µg/kg, 1 x 4-6 iv.) and maintaining normovolaemia;
  * Reduction of mean arterial pressure and neuroprotection with Nimodipine infusion 5 ml per hour for 21 days and Urapidil 200 mg /200 ml, 7-10 ml/h.
  * Control of ICP, which can be in majority of patients, kept at values below 15 mmHg.
  Arms: Intracranial pressure-targeted therapy
Procedure: Cerebral perfusion pressure-targeted therapy — * ICP monitoring using an external ventricular drain and CSF drainage as a first measure if ICP was increased (over 15-20 mmHg);
  * Maintenance of CPP over 70-80 mmHg (Triple 'H' therapy = 3L/24 hours including 1L of colloids - 5% albumin; drugs = dopamine, dobutamine);
  * No hyperventilation if ICP was under 20-25 mmHg and hyperventilation as a third measure if ICP was increased;
  * Osmotherapy (20% manitol, bolus 150-350 ml or 10% manitol, 50 ml/h for 10 hours and standard electrolytes [Na, Cl and K]);
  Arms: Cerebral perfusion pressure-targeted

SUMMARY:
Secondary brain ischaemia (SBI) usually develops after aneurysmal subarachnoid haemorrhage (SAH) and severe traumatic brain injury (TBI). The current management strategies are based on intracranial pressure-targeted therapy (ICP-targeted) with cerebral microdialysis monitoring (modified Lund concept) or cerebral perfusion pressure-targeted therapy (CPP-targeted). We present a randomised controlled study to compare the two management strategies.

The hypotheses of the study were:

* SBI developed after aneurysmal SAH and severe TBI share the same crucial characteristics and any treatment applied will essentially treat the same underlying pathophysiology.
* ICP-targeted therapy with cerebral microdialysis monitoring according to the modified Lund concept is superior to CPP-targeted therapy in managing comatose patients with SBI after aneurysmal SAH and severe TBI.

Sixty comatose operated patients with SBI following aneurysmal SAH and severe TBI were randomized into ICP-targeted therapy with cerebral microdialysis monitoring and CPP-targeted therapy groups. Mortality rates in both groups were calculated and biochemical signs of cerebral ischaemia were analysed using cerebral microdialysis. Outcome for cerebral microdialysis was measured as poor outcome (Glasgow Outcome Scale score 1, 2 and 3) or good outcome (Glasgow Outcome Scale score 4 and 5).

ELIGIBILITY:
Inclusion Criteria:

* patients with subarachnoid haemorrhage who had anterior circulation aneurysm rupture only
* multiple anterior aneurysm rupture
* severe traumatic brain injury with isolated head injury and intradural focal lesions only

Exclusion Criteria:

* Glasgow Outcome Score of 3 with or without brainstem reflexes
* Significant co-morbidities
* posterior circulation aneurysm
* multisystem injuries
* diffuse axonal injuries

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 18 months
  Measurement of outcome was done using the Glasgow Outcome Scale (GOS) after each specific intervention in all the patients. GOS 1 - dead, 2- vegetative, 3- severe disabled, 4- moderate disabled, 5- independent.

CONTACTS AND LOCATIONS:
Overall Officials: Kemal Dizdarevic, MD, MSc, PhD, Principal Investigator — Department of Neurosurgery, Clinical Centre University of Sarajevo, Sarajevo, Bosnia and Herzegovina
Locations (1):
- Department of Neurosurgery, Clinical Centre University of Sarajevo, Sarajevo, Bosnia and Herzegovina